CLINICAL TRIAL: NCT05750563
Title: Randomised, Double-blind, Placebo-controlled, Parallel-group, Multicentre, Interventional Clinical Trial to Assess the Efficacy and Safety of the Food Supplement Microsmin® Plus in the Symptomatic Treatment of Haemorrhoids
Brief Title: Randomised, Double-blind, Placebo-controlled to Assess the Efficacy and Safety of the Food Supplement Microsmin® Plus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Giellepi S.p.A (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPGIE/0122/FS
Record Dates: First submitted 2023-02-14; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Haemorrhoids
Keywords: haemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Diosmin

STUDY DESIGN:
Intervention Model Description: DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP OF THE FOOD SUPPLEMENT MICROSMIN® PLUS (DIOSMIN AND MICRONIZED FLAVONOIDS)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Investigational food supplement placebo will be administered according to the same schedule provided for the active product:
  * From day 1 to day 4: 1 tablet three times a day, before meals (breakfast, lunch and dinner)
  * From day 5 to day 7: 1 tablet twice a day, before breakfast and dinner
  * From day 8 to day 62: 1 tablet once a day, before breakfast
  Interventions: Other: Placebo
- Experimental (Experimental): The dosage will be the following:
  * From day 1 to day 4: 1 tablet three times a day, before meals (breakfast, lunch and dinner)
  * From day 5 to day 7: 1 tablet twice a day, before breakfast and dinner
  * From day 8 to day 62: 1 tablet once a day, before breakfast
  Interventions: Dietary Supplement: diosmin and micronized flavonoids

INTERVENTIONS:
Dietary Supplement: diosmin and micronized flavonoids — the symptomatic treatment of haemorrhoids
  Other Names: MICROSMIN® PLUS
  Arms: Experimental
Other: Placebo — Use as comparator
  Arms: Placebo

SUMMARY:
Haemorrhoids are variceal dilatations of the anal and perianal venous plexus and often develop secondary to the persistently elevated venous pressure within the haemorrhoidal plexus .

The classical position of haemorrhoids corresponds to three positions which are the right anterior, right posterior and the left lateral areas of the anal canal. Haemorrhoids may be external or internal. External haemorrhoids are covered with skin and internal haemorrhoids are covered with anal mucous membranes. The grading system used by Banov to classify internal haemorrhoids is one of the most common grading systems used by clinicians and is used to guide therapeutic practice. Internal haemorrhoids can be divided into four categories depending on the degree of prolapse (the protrusion of the haemorrhoid through the anus). The most widely accepted classification is the Goligher classification:

* Bleeding but no prolapse (grade I).
* Hemorrhoidal piles prolapse through the anus during straining, but they reduce spontaneously (grade II).
* Hemorrhoidal piles prolapse through the anus during straining and require manual reduction (grade III).
* The prolapse is irreducible (grade IV). Most symptoms and signs which patients present with arise from internal haemorrhoids, derive from structural changes of the normal anatomic padding (enlarged internal haemorrhoids) and are generally associated with chronic straining either due to constipation, diarrhoea or prolonged periods trying to defecate. They are also common during pregnancy and childbirth.

DETAILED DESCRIPTION:
Haemorrhoids are variceal dilatations of the anal and perianal venous plexus and often develop secondary to the persistently elevated venous pressure within the haemorrhoidal plexus .

The classical position of haemorrhoids corresponds to three positions which are the right anterior, right posterior and the left lateral areas of the anal canal. Haemorrhoids may be external or internal. External haemorrhoids are covered with skin and internal haemorrhoids are covered with anal mucous membranes. The grading system used by Banov to classify internal haemorrhoids is one of the most common grading systems used by clinicians and is used to guide therapeutic practice. Internal haemorrhoids can be divided into four categories depending on the degree of prolapse (the protrusion of the haemorrhoid through the anus). The most widely accepted classification is the Goligher classification :

* Bleeding but no prolapse (grade I).
* Hemorrhoidal piles prolapse through the anus during straining, but they reduce spontaneously (grade II).
* Hemorrhoidal piles prolapse through the anus during straining and require manual reduction (grade III).
* The prolapse is irreducible (grade IV). Most symptoms and signs which patients present with arise from internal haemorrhoids, derive from structural changes of the normal anatomic padding (enlarged internal haemorrhoids) and are generally associated with chronic straining either due to constipation, diarrhoea or prolonged periods trying to defecate. They are also common during pregnancy and childbirth.

The acute clinical manifestation of the hemorrhoidal disease (commonly known as "hemorrhoidal crisis") is characterized by symptoms and signs, also common in chronic pathologies, such as rectal bleeding, prolapse, pruritus (itching), pain, oedema, often thrombosis, and less frequently soiling or mucoid discharge. Rectal bleeding (the most common presenting sign) is classically bright red as there is a high blood oxygen content within the arteriovenous anastomosis. This bleeding is usually described as bright red spotting on the toilet tissue or dripping in the toilet bowl and normally occurs at the end of defecation, separately from the stool. External haemorrhoids may be asymptomatic or associated with discomfort or with acute extreme pain in the event of a local thrombosis (formation of a clot).

Phlebotonics are a heterogenous class of drugs consisting of plant extracts (i.e., flavonoids) and synthetic compounds. Although their precise mechanism of action has not been fully established, they are known to strengthen blood vessel walls, improve venous tone, stabilise capillary permeability and increase lymphatic drainage. They have been used to treat a variety of conditions including chronic venous insufficiency, lymphoedema and haemorrhoids. In particular, numerous trials assessing the effect of phlebotonics in treating the symptoms and signs of haemorrhoidal disease (they are generally used in the less severe stages of haemorrhoids, first and second-grade haemorrhoids and during the thrombosis episodes) suggest that there is a potential benefit. Moreover, 2 reviews and 1 systematic review evaluated the micronized purified flavonoid fraction (MPFF) activities and performance in haemorrhoids.

Based on the available clinical evidence, current national guidelines and extensive clinical experience in treating patients affected by the haemorrhoidal disease, MPFF can be administered as a first-line treatment, in combination with diet (increased fibre and fluid intake) and lifestyle modifications, for acute grade I/II HD.

A new micronized formulation of diosmin was incorporated in a new dietary supplement called Microsmin® Plus to increase plasma concentrations due to the property manufacturing process able to improve intestinal absorption following oral intake. This product has evidenced a better bioavailability compared with micronized diosmin in rats (4-fold increased) and in healthy volunteers (19) (9.4 greater with higher plasmatic concentrations).

Moreover, a randomized, double-blind, placebo-controlled trial carried out in patients with chronic venous disease (CVD) showed that the administration of a low dose of Microsmin® Plus is safe and effective in relieving symptoms and improving QoL in patients with CVD after 8 weeks of treatment.

This study aims to investigate the efficacy and safety of phlebotonics (dietary supplement containing micronized diosmin, i.e., Microsmin® Plus) in alleviating the signs, symptoms and severity of haemorrhoidal disease in a set of standard clinical practices where the administration of phlebotonics is integrated with lifestyle counselling. Therefore, the Research Question of the present trial is the following: in a population of adult patients, men and women, suffering from symptomatic haemorrhoids, will the administration of the dietary supplement Microsmin® Plus (diosmin and micronized flavonoids) for 63 days (7-days acute treatment phase + 55-days maintenance phase), integrated with lifestyle counselling, improve the symptomatology (clinical signs and symptoms) in comparison with patients receiving placebo, results observed after 4, 7 and 63 days after the beginning of the treatment?

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥ 18 and ≤ 60 years. The sex will be balanced by randomized stratification.
2. Patients diagnosed with Grade I - II symptomatic haemorrhoids (according to Goligher classification) confirmed by clinical and anoscopic or proctoscopic examination performed within 3 months before baseline. Ultrasound examination at baseline is recommended, but not mandatory.
3. Patient free from the following treatments for haemorrhoids from at least 4 weeks: laser treatments for haemorrhoids, steroidal or non-steroidal anti-inflammatory drugs, analgesics (other than the rescue medicine indicated in the protocol), any anti-hemorrhoidal treatment (included phlebotonic compounds both drugs and dietary supplements), anticoagulants, and antiplatelet agents.
4. Able to communicate adequately with the Investigator and to comply with the requirements for the entire study.
5. Capable of and freely willing to provide written informed consent prior to participating in the study.

Exclusion Criteria:

1. Inflammatory and infectious disease of the digestive tract (e.g., IBD - Inflammatory Bowel Diseases).
2. Acute haemorrhoids or complicated haemorrhoids with bleeding requiring admission, such as strangulated internal haemorrhoids, thrombosed internal or external haemorrhoids.
3. Previous haemorrhoidectomy or previous laser treatment.
4. Moderate to severe hypertension, cardiovascular diseases, renal failure, cirrhosis, colorectal cancer, anal fissure or fistula.
5. Use of laser treatments for haemorrhoids, steroidal or non-steroidal anti-inflammatory drugs, analgesics (other than the rescue medicine indicated in the protocol), any anti-hemorrhoidal treatment (included phlebotonic compounds both drugs and dietary supplements), anticoagulants, and antiplatelet agents in the 4 weeks prior to inclusion and during the whole study.
6. Alcohol or drug abuse.
7. Patients considered smokers (≥10 cigarettes/day).
8. Energy-restricted diet for weight loss.
9. Pregnant woman, lactating woman, and woman of childbearing potential who is planning a pregnancy or is unwilling to use appropriate methods of contraception* during the study.

   *Methods of contraception: hormonal contraceptive, intrauterine device or intrauterine system, double barrier method (condom with spermicide/diaphragm or cervical cap with spermicide), surgical sterilization (vasectomy, tubal ligation, etc.).
10. Hypersensitivity to active principle (diosmin) or to any other ingredient contained in the tested food supplement.
11. History of anaphylaxis or severe complicated allergy symptoms.
12. Patients unlikely to cooperate.
13. Patients with any other medical condition that, in the opinion of the Investigator, would compromise participation or be likely to lead to hospitalisation during the study.
14. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of the tested food supplement Microsmin® Plus | 63 days
  Evaluate the efficacy of the tested food supplement Microsmin® Plus (diosmin and micronized flavonoids) in comparison with placebo in the symptomatic treatment of haemorrhoids in adult patients affected by Grade I-II (Goligher classification) haemorrhoids as assessed by the patient at the end of the treatment period.
To evaluate the safety of the tested food supplement through adverse events and serious adverse events incidence assessed by Investigators and reported according to the current legislation | 63 days
  To evaluate the safety of the tested food supplement through AE and SAE incidence assessed by Investigators and reported according to the current legislation.

SECONDARY OUTCOMES:
To evaluate the early efficacy of the tested food supplement in comparison with placebo in the symptomatic treatment of haemorrhoids as assessed by the patient after 4 and 7 days of treatment | 63 days
  To evaluate the early efficacy of the tested food supplement in comparison with placebo in the symptomatic treatment of haemorrhoids as assessed by the patient after 4 and 7 days of treatment.
To evaluate the efficacy of the tested food supplement in comparison with placebo in the clinical improvement of haemorrhoids as assessed by the Investigator at each visit (day 7 and 63) | 63 days
  To evaluate the efficacy of the tested food supplement in comparison with placebo in the clinical improvement of haemorrhoids as assessed by the Investigator at each visit (days 7 and 63).
To evaluate analgesic consumption in patients treated with the tested food supplement in comparison with placebo as reported by the patient in the diary | 63 days
  To evaluate analgesic consumption in patients treated with the tested food supplement in comparison with placebo as reported by the patient in the diary.
To assess the overall satisfaction with the tested food supplement in comparison with placebo according to patient's judgement, at the end of the treatment period (day 63) | 63 days
  To assess the overall satisfaction with the tested food supplement in comparison with placebo according to patient's judgement, at the end of the treatment period (day 63).
To assess the improvement in the quality of life by means of the Short Heath Scale for Hemorrhoidal Disease (SHSHD) score; assessed by patients after 7 and 63 days of treatment | 63 days
  To assess the improvement in the quality of life by means of the Short Heath Scale for Hemorrhoidal Disease (SHSHD) score; assessed by patients after 7 and 63 days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Terruzzi, CSO, Study Director — Giellepi S.p.A
Locations (1):
- SC Salvosan Ciobanca SRL, Zalău, Sălaj County, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lohsiriwat V. Hemorrhoids: from basic pathophysiology to clinical management. World J Gastroenterol. 2012 May 7;18(17):2009-17. doi: 10.3748/wjg.v18.i17.2009. PMID 22563187
- [Background] Sanchez C, Chinn BT. Hemorrhoids. Clin Colon Rectal Surg. 2011 Mar;24(1):5-13. doi: 10.1055/s-0031-1272818. PMID 22379400
- [Background] Banov L Jr, Knoepp LF Jr, Erdman LH, Alia RT. Management of hemorrhoidal disease. J S C Med Assoc. 1985 Jul;81(7):398-401. No abstract available. PMID 3861909
- [Background] Thomson JPS, Goligher JC. Surgery of the anus, rectum and colon. J. C. Goligher. Fourth Edition. 264 × 198 mm. Pp. 968 + vii, with 654 illustrations. 1980. London: Baillière Tindall. £35·00. BJS Br J Surg. 1980;67(7):532-532
- [Background] Rubbini M, Ascanelli S. Classification and guidelines of hemorrhoidal disease: Present and future. World J Gastrointest Surg. 2019 Mar 27;11(3):117-121. doi: 10.4240/wjgs.v11.i3.117. PMID 31057696
- [Background] Perera N, Liolitsa D, Iype S, Croxford A, Yassin M, Lang P, Ukaegbu O, van Issum C. Phlebotonics for haemorrhoids. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD004322. doi: 10.1002/14651858.CD004322.pub3. PMID 22895941
- [Background] Colak T, Akca T, Dirlik M, Kanik A, Dag A, Aydin S. Micronized flavonoids in pain control after hemorrhoidectomy: a prospective randomized controlled study. Surg Today. 2003;33(11):828-32. doi: 10.1007/s00595-003-2604-5. PMID 14605954
- [Background] La Torre F, Nicolai AP. Clinical use of micronized purified flavonoid fraction for treatment of symptoms after hemorrhoidectomy: results of a randomized, controlled, clinical trial. Dis Colon Rectum. 2004 May;47(5):704-10. doi: 10.1007/s10350-003-0119-1. Epub 2004 Mar 25. PMID 15037936
- [Background] Corsale I, Carrieri P, Martellucci J, Piccolomini A, Verre L, Rigutini M, Panicucci S. Flavonoid mixture (diosmin, troxerutin, rutin, hesperidin, quercetin) in the treatment of I-III degree hemorroidal disease: a double-blind multicenter prospective comparative study. Int J Colorectal Dis. 2018 Nov;33(11):1595-1600. doi: 10.1007/s00384-018-3102-y. Epub 2018 Jun 22. PMID 29934701
- [Background] Cospite M. Double-blind, placebo-controlled evaluation of clinical activity and safety of Daflon 500 mg in the treatment of acute hemorrhoids. Angiology. 1994 Jun;45(6 Pt 2):566-73. PMID 8203789
- [Background] Giannini I, Amato A, Basso L, Tricomi N, Marranci M, Pecorella G, Tafuri S, Pennisi D, Altomare DF. Flavonoids mixture (diosmin, troxerutin, hesperidin) in the treatment of acute hemorrhoidal disease: a prospective, randomized, triple-blind, controlled trial. Tech Coloproctol. 2015 Jun;19(6):339-45. doi: 10.1007/s10151-015-1302-9. Epub 2015 Apr 19. PMID 25893991
- [Background] Giannini I, Amato A, Basso L, Tricomi N, Marranci M, Pecorella G, Tafuri S, Pennisi D, Altomare DF. Erratum to: Flavonoids mixture (diosmin, troxerutin, hesperidin) in the treatment of acute hemorrhoidal disease: a prospective, randomized, triple-blind, controlled trial. Tech Coloproctol. 2015 Oct;19(10):665-6. doi: 10.1007/s10151-015-1357-7. No abstract available. PMID 26338366
- [Background] Jiang ZM, Cao JD. The impact of micronized purified flavonoid fraction on the treatment of acute haemorrhoidal episodes. Curr Med Res Opin. 2006 Jun;22(6):1141-7. doi: 10.1185/030079906X104803. PMID 16846547
- [Background] Lyseng-Williamson KA, Perry CM. Micronised purified flavonoid fraction: a review of its use in chronic venous insufficiency, venous ulcers and haemorrhoids. Drugs. 2003;63(1):71-100. doi: 10.2165/00003495-200363010-00005. PMID 12487623
- [Background] La Torre F, Nicolai AP, Otti M. [Hemorrhoids and conservative treatment. Review of the literature on the use of diosmin and micronized hesperidin]. Minerva Chir. 1999 Dec;54(12):909-16. No abstract available. Italian. PMID 10736998
- [Background] Sheikh P, Lohsiriwat V, Shelygin Y. Micronized Purified Flavonoid Fraction in Hemorrhoid Disease: A Systematic Review and Meta-Analysis. Adv Ther. 2020 Jun;37(6):2792-2812. doi: 10.1007/s12325-020-01353-7. Epub 2020 May 12. PMID 32399811
- [Background] Godeberge P, Sheikh P, Lohsiriwat V, Jalife A, Shelygin Y. Micronized purified flavonoid fraction in the treatment of hemorrhoidal disease. J Comp Eff Res. 2021 Jul;10(10):801-813. doi: 10.2217/cer-2021-0038. Epub 2021 Apr 30. PMID 33928786
- [Background] Russo R, Mancinelli A, Ciccone M, Terruzzi F, Pisano C, Severino L. Pharmacokinetic Profile of microSMIN Plus, a new Micronized Diosmin Formulation, after Oral Administration in Rats. Nat Prod Commun. 2015 Sep;10(9):1569-72. PMID 26594761
- [Background] Russo R, Chandradhara D, De Tommasi N. Comparative Bioavailability of Two Diosmin Formulations after Oral Administration to Healthy Volunteers. Molecules. 2018 Aug 29;23(9):2174. doi: 10.3390/molecules23092174. PMID 30158431
- [Background] Serra R, Ielapi N, Bitonti A, Candido S, Fregola S, Gallo A, Loria A, Muraca L, Raimondo L, Velcean L, Guadagna S, Gallelli L. Efficacy of a Low-Dose Diosmin Therapy on Improving Symptoms and Quality of Life in Patients with Chronic Venous Disease: Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2021 Mar 19;13(3):999. doi: 10.3390/nu13030999. PMID 33808784
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Sun Z, Migaly J. Review of Hemorrhoid Disease: Presentation and Management. Clin Colon Rectal Surg. 2016 Mar;29(1):22-9. doi: 10.1055/s-0035-1568144. PMID 26929748
- [Background] Everhart JE, Ruhl CE. Burden of digestive diseases in the United States part I: overall and upper gastrointestinal diseases. Gastroenterology. 2009 Feb;136(2):376-86. doi: 10.1053/j.gastro.2008.12.015. Epub 2009 Jan 3. No abstract available. PMID 19124023
- [Background] Ganz RA. The evaluation and treatment of hemorrhoids: a guide for the gastroenterologist. Clin Gastroenterol Hepatol. 2013 Jun;11(6):593-603. doi: 10.1016/j.cgh.2012.12.020. Epub 2013 Jan 16. No abstract available. PMID 23333220
- [Background] Heaton ND, Davenport M, Howard ER. Symptomatic hemorrhoids and anorectal varices in children with portal hypertension. J Pediatr Surg. 1992 Jul;27(7):833-5. doi: 10.1016/0022-3468(92)90377-j. PMID 1640328
- [Background] Johanson JF, Sonnenberg A. The prevalence of hemorrhoids and chronic constipation. An epidemiologic study. Gastroenterology. 1990 Feb;98(2):380-6. doi: 10.1016/0016-5085(90)90828-o. PMID 2295392
- [Background] Szyca R, Leksowski K. Assessment of patients' quality of life after haemorrhoidectomy using the LigaSure device. Wideochir Inne Tech Maloinwazyjne. 2015 Apr;10(1):68-72. doi: 10.5114/wiitm.2015.49672. Epub 2015 Mar 10. PMID 25960796
- [Background] Tjandra JJ, Tan JJ, Lim JF, Murray-Green C, Kennedy ML, Lubowski DZ. Rectogesic (glyceryl trinitrate 0.2%) ointment relieves symptoms of haemorrhoids associated with high resting anal canal pressures. Colorectal Dis. 2007 Jun;9(5):457-63. doi: 10.1111/j.1463-1318.2006.01134.x. PMID 17504344
- [Background] Lichota A, Gwozdzinski L, Gwozdzinski K. Therapeutic potential of natural compounds in inflammation and chronic venous insufficiency. Eur J Med Chem. 2019 Aug 15;176:68-91. doi: 10.1016/j.ejmech.2019.04.075. Epub 2019 May 6. PMID 31096120
- [Background] Lebeau J, Furman C, Bernier JL, Duriez P, Teissier E, Cotelle N. Antioxidant properties of di-tert-butylhydroxylated flavonoids. Free Radic Biol Med. 2000 Nov 1;29(9):900-12. doi: 10.1016/s0891-5849(00)00390-7. PMID 11063915
- [Background] Panche AN, Diwan AD, Chandra SR. Flavonoids: an overview. J Nutr Sci. 2016 Dec 29;5:e47. doi: 10.1017/jns.2016.41. eCollection 2016. PMID 28620474
- [Background] Durga M. International Journal of Pharma and Bio Sciences MULTIFARIOUS ACTIONS OF DIETARY FLAVONOIDS IMPLICATIONS IN CANCER AND CATARACT ABSTRACT [Internet]. kipdf.com. [cited 2022 Jun 24]. Available from: https://kipdf.com/international-journal-of-pharma-and-bio-sciences-multifarious-actions-of-dietary_5ada41157f8b9a2e7e8b45c7.html
- [Background] Rabe E, Guex JJ, Morrison N, Ramelet AA, Schuller-Petrovic S, Scuderi A, Staelens I, Pannier F. Treatment of chronic venous disease with flavonoids: recommendations for treatment and further studies. Phlebology. 2013 Sep;28(6):308-19. doi: 10.1177/0268355512471929. Epub 2013 May 6. PMID 23395842
- [Background] Monograph. Diosmin. Altern Med Rev. 2004 Sep;9(3):308-11. No abstract available. PMID 15387721
- [Background] Snow G. blockrand: Randomization for Block Random Clinical Trials [Internet]. 2020 [cited 2022 Jun 9]. Available from: https://CRAN.R-project.org/package=blockrand
- [Background] Uschner D, Schindler D, Hilgers RD, Heussen N. randomizeR : An R Package for the Assessment and Implementation of Randomization in Clinical Trials. J Stat Softw [Internet]. 2018 [cited 2022 Jun 9];85(8). Available from: http://www.jstatsoft.org/v85/i08/
- [Background] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604
- [Background] Slappendel R, Simpson K, Dubois D, Keininger DL. Validation of the PAC-SYM questionnaire for opioid-induced constipation in patients with chronic low back pain. Eur J Pain. 2006 Apr;10(3):209-17. doi: 10.1016/j.ejpain.2005.03.008. PMID 15914049
- [Background] Hjortswang H, Jarnerot G, Curman B, Sandberg-Gertzen H, Tysk C, Blomberg B, Almer S, Strom M. The Short Health Scale: a valid measure of subjective health in ulcerative colitis. Scand J Gastroenterol. 2006 Oct;41(10):1196-203. doi: 10.1080/00365520600610618. PMID 16990205
- [Background] Stjernman H, Granno C, Jarnerot G, Ockander L, Tysk C, Blomberg B, Strom M, Hjortswang H. Short health scale: a valid, reliable, and responsive instrument for subjective health assessment in Crohn's disease. Inflamm Bowel Dis. 2008 Jan;14(1):47-52. doi: 10.1002/ibd.20255. PMID 17828783
- [Background] Rorvik HD, Styr K, Ilum L, McKinstry GL, Dragesund T, Campos AH, Brandstrup B, Olaison G. Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum. 2019 Mar;62(3):333-342. doi: 10.1097/DCR.0000000000001234. PMID 30451751
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830